CLINICAL TRIAL: NCT06058442
Title: The Pancreatic Enzymes After Gastrectomy Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Albrecht Hoffmeister, Prof. Dr. med., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PANEM
Record Dates: First submitted 2023-09-08; First posted 2023-09-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Gastrectomy
Keywords: enzyme supplementation; lipase; elastase; gastrointestinal; quality of life
MeSH Terms: interventions — nortase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NORTASE® (Experimental)
  Interventions: Drug: NORTASE®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NORTASE® — 10-15 capsules of NORTASE® per day - over 6 months
  Arms: NORTASE®
Drug: Placebo — 10-15 capsules of placebo per day - over 6 months
  Arms: Placebo

SUMMARY:
This trial evaluates the effects (e.g. on quality of life, weight) of NORTASE® compared to standard care of patients who have undergone gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Gastrectomy (total and partial); at least > 50 % of the stomach must be resected
2. Age 18 or older
3. Written informed consent

Exclusion Criteria:

1. Indication for pancreas enzyme therapy
2. Gastrectomy with palliative intention
3. UICC (Union for International Cancer Control) Stage IV gastric malignancy
4. Malnutrition of other aetiology
5. Life expectancy < 12 months
6. Known lactose intolerance
7. Known hereditary galactose intolerance
8. Patients on alpha-glucosidase inhibitors (AGIs)
9. Acute pancreatitis
10. Acute episode of chronic pancreatitis
11. Known hypersensitivity to moulds (mould allergy) or any other ingredient of NORTASE®
12. Participation in competing interventional trials may be allowed under circumstances
13. Patients under legal supervision or guardianship
14. Patients who are dependent on the investigator or the medical staff of the trial team or the coordinating investigator or the sponsor
15. Fertile women (within two years of their last menstruation) without appropriate contraceptive measures (implanon, injections, oral contraceptives, intrauterine devices, partner with vasectomy) while participating in the trial
16. Pregnant or nursing women
17. Suspected lack of compliance
18. Patients who were already enrolled in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Disease specific quality of life (QOL) | 6 months
  This is the physical sub-score from the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC-QLQ-C30) and ranges from 0 (lowest physical functioning) to 100 (highest physical functioning).

SECONDARY OUTCOMES:
Nutritional supplementation or weight loss | 6 months
  Proportion of patients who receive supplemental nutrition after the run-in period of 3 weeks or have > 10% weight loss at six months
Weight | 6 months
  Percent weight-change at six months (weight in kilograms)
Serum haemoglobin | 6 months
  Concentration of serum haemoglobin
Total protein | 6 months
  Concentration of total protein
Albumin | 6 months
  Concentration of albumin
Glucose | 6 months
  Concentration of glucose
HbA1c | 6 months
  Concentration of HbA1c
Cholesterol | 6 months
  Concentration of cholesterol
Vitamin A | 6 months
  Concentration of vitamin A
Vitamin B12 | 6 months
  Concentration of vitamin B12
Vitamin D | 6 months
  Concentration of vitamin D
Vitamin E | 6 months
  Concentration of vitamin E
Vitamin K | 6 months
  Concentration of vitamin K

OTHER OUTCOMES:
Faecal elastase-1 | 6 months
  Concentration of faecal elastase-1

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Hoffmeister, Prof. Dr., Principal Investigator — Universität Leipzig
Locations (9):
- Germany (9):
  - Sana Kliniken Leipziger Land GmbH, Klinik für Allgemein-, Viszeral-, MIC- und Gefäßchirurgie / Thoraxchirurgie, Borna
  - Carl-Thiem-Klinikum Cottbus gGmbH; 4. Medizinische Klinik, Cottbus
  - KEM | Evang. Kliniken Essen-Mitte gGmbH, Klinik für Internistische Onkologie, Essen
  - UNIVERSITÄTSKLINIKUM FREIBURG Klinik für Allgemein- und Viszeralchirurgie Department Chirurgie, Freiburg im Breisgau
  - Universitätsklinikum Jena, Allgemein-, Viszeral- und Gefäßchirurgie, Jena
  - Klinik und Poliklinik für Onkologie, Gastroenterologie, Hepatologie und Pneumologie Universitätsklinikum Leipzig, Leipzig
  - Klinikum St. Georg, Abteilung für Allgemein-, Viszeral- und Onkologische Chirurgie, Leipzig
  - Helios Kliniken Schwerin; Klinik für Allgemein- und Viszeralchirurgie, Schwerin
  - Klinik für Allgemein- und Viszeralchirurgie, Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided